CLINICAL TRIAL: NCT05672771
Title: The Effects of Mixed Working Memory Training on Subsequent Training Gains Among Older Adults
Acronym: MixedWM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Elizabeth A L Stine-Morrow, Professor Emerita, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Mixed Working Memory Training; R56AG058708 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2023-01-05 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cognitive Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Different Mixed Condition (DM) (Experimental): Training in both Lexical Decision Span and Category Span in Phase 1 (which are both different from the target task Reading Span in Phase 2).
  Interventions: Behavioral: Different Mixed Condition (DM)
- Different Single Condition (DS) (Experimental): Training in the Lexical Decision Span in Phase 1 (which is different from the target task Reading Span in Phase 2).
  Interventions: Behavioral: Different Single Condition (DS)
- Same Task (ST) Practice Control (Active Comparator): Training in Reading Span task in Phase 1 (which is the same as target task in Phase 2).
  Interventions: Behavioral: Same Task (ST) Practice Control
- Non-WM Placebo Control (PC) (Placebo Comparator): Training in a speeded Lexical Decision task only (which has no memory component) in Phase 1 prior to Phase 2 training in WM.
  Interventions: Behavioral: Non-WM Placebo Control (PC)

INTERVENTIONS:
Behavioral: Different Mixed Condition (DM) — Participants engage in home-based training on two working memory tasks, both different from those in the target task training. Goal is 10 days of training, with 4 8-min blocks of training each day.
  Arms: Different Mixed Condition (DM)
Behavioral: Different Single Condition (DS) — Participants engage in home-based training on a working memory task that is different from that in the target task training. Goal is 10 days of training, with 4 8-min blocks of training each day.
  Arms: Different Single Condition (DS)
Behavioral: Same Task (ST) Practice Control — Participants engage in home-based training on the exact same working memory tasks as that in the target task training. Goal is 10 days of training, with 4 8-min blocks of training each day.
  Arms: Same Task (ST) Practice Control
Behavioral: Non-WM Placebo Control (PC) — Participants engage in home-based training on speeded verbal decision, which unlike the target task training, has no memory component. Goal is 10 days of training, with 4 8-min blocks of training each day.
  Arms: Non-WM Placebo Control (PC)

SUMMARY:
While an intellectually active and socially integrated lifestyle shows promise for promoting cognitive resilience, the mechanisms underlying any such effects are not well understood. The aim of the current project is test the implications of the "mutualism" hypothesis, which suggests that intellectual function emerges out of the reciprocal influence of growth in abilities as they are exercised in the ecology of everyday life. Such a view implies that improvement in one component will enhance the modifiability of a related component. An additional aim was to test the idea that mutualistic effects will be enhanced by more diverse training in related skills, such as interleaved training of multiple skills, relative to single-component training.

A "successive-enrichment" paradigm was developed to test this with working memory (WM) as the target for training given its centrality in models of attention, intellectual function, and everyday capacities such as reasoning and language comprehension. All participants receive the same target training, but the nature of the training that precedes it is manipulated. Outcome measures include pre- to posttest gains in working memory and episodic memory, as well as the rate of gain in learning the target task. The principle of enhanced mutualism would predict that more diverse experiences related to the target skill will enhance efficiency in acquiring the target skill.

DETAILED DESCRIPTION:
Within conventional assessments of transfer that examine the effects of training on measures of function at a single time point, these ideas has not been tested. In this project, a "successive-enrichment" paradigm was used to examine improvement in cognitive skills as a function of different conditions for earlier training. The target for training is working memory (WM) given its centrality in models of attention, intellectual function, and everyday capacities such as reasoning and language comprehension.

In the successive-enrichment paradigm, all participants receive the same target training, but the nature of the training that precedes it is manipulated. Thus, in Phase 2, all participants are trained for 10 days on the reading span task (RdgS), in which the task is to verify sensibility in a set of sentences and retain in memory an alphabetic character presented after each sentence. The set size adapts to the participant's skill (in both accuracy of sensibility decisions and memory for the letter set). In Phase 1, participants are randomly assigned to one of four groups designed to test the assumption that related and diverse experiences with the target skill differentially enhance the rate of learning the new skill. In the Same Task (ST) control, participants train on the RdgS, and were expected to be at ceiling in Phase 2. In the Different Single condition (DS), participants trained on a WM task different from that in Phase 1 (the lexical decision span). In the Different Mixed (DM) condition, participants trained on two different interleaved WM tasks, the lexical decision span and the category span. In the non-WM Placebo Control (PC), participants train on a speeded lexical decision task (matched in materials and verbal decision component to the lexical decision span the but requiring no simultaneous memory.

Outcome measures include pre- to posttest gains in working memory and episodic memory, as well as the rate of gain in learning the RdgS in Phase 2. The PC and ST controls define the lower and upper limits of performance, respectively. The principle of enhanced mutualism would predict that the DM group will show more efficient learning of the RdgS in Phase 2 than the DS group, which will both show more efficient learning than the PC group.

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers or acquisition of English before age 6 yrs old
* Self-report of hearing ability sufficient to engage with lab personnel
* No stroke in the last 3 years
* No current cancer treatment involving radiation or chemotherapy - No self-reported learning disability
* No self-reported psychiatric disorder
* Willingness to be randomly assigned to training conditions
* No plans that would limit participation during the activity period
* No participation in a cognitive intervention program in the last year

No additional Exclusion Criteria.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A L Stine-Morrow, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Beckman Institute, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data and Analytic Code will be made available on OSF.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After completion and paper is published (~2025)

REFERENCES:
- [Background] Stine-Morrow EAL, Payne BR, Roberts BW, Kramer AF, Morrow DG, Payne L, Hill PL, Jackson JJ, Gao X, Noh SR, Janke MC, Parisi JM. Training versus engagement as paths to cognitive enrichment with aging. Psychol Aging. 2014 Dec;29(4):891-906. doi: 10.1037/a0038244. Epub 2014 Nov 17. PMID 25402337
- [Background] Payne BR, Stine-Morrow EAL. The Effects of Home-Based Cognitive Training on Verbal Working Memory and Language Comprehension in Older Adulthood. Front Aging Neurosci. 2017 Aug 8;9:256. doi: 10.3389/fnagi.2017.00256. eCollection 2017. PMID 28848421
- [Background] Savi AO, Marsman M, van der Maas HLJ, Maris GKJ. The Wiring of Intelligence. Perspect Psychol Sci. 2019 Nov;14(6):1034-1061. doi: 10.1177/1745691619866447. Epub 2019 Oct 24. PMID 31647746
- [Background] van der Maas HL, Dolan CV, Grasman RP, Wicherts JM, Huizenga HM, Raijmakers ME. A dynamical model of general intelligence: the positive manifold of intelligence by mutualism. Psychol Rev. 2006 Oct;113(4):842-61. doi: 10.1037/0033-295X.113.4.842. PMID 17014305
- [Background] Van Der Maas HLJ, Kan KJ, Marsman M, Stevenson CE. Network Models for Cognitive Development and Intelligence. J Intell. 2017 Apr 20;5(2):16. doi: 10.3390/jintelligence5020016. PMID 31162407
- [Background] Daneman M, Merikle PM. Working memory and language comprehension: A meta-analysis. Psychon Bull Rev. 1996 Dec;3(4):422-33. doi: 10.3758/BF03214546. PMID 24213976
- [Background] Stine-Morrow, E. A. L., & Manavbasi, I. (2022). Beyond "Use It or Lose It": The impact of engagement on cognitive aging. Annual Review of Developmental Psychology, 4, 319-352.
- [Background] Brown, P. C., Roediger, H. L., & McDaniel, M. A. (2014). Make it stick: The science of successful learning. Harvard University Press.
- [Background] Engle RW, Tuholski SW, Laughlin JE, Conway ARA. Working memory, short-term memory, and general fluid intelligence: a latent-variable approach. J Exp Psychol Gen. 1999 Sep;128(3):309-331. doi: 10.1037//0096-3445.128.3.309. PMID 10513398
- [Result] Conway AR, Kane MJ, Bunting MF, Hambrick DZ, Wilhelm O, Engle RW. Working memory span tasks: A methodological review and user's guide. Psychon Bull Rev. 2005 Oct;12(5):769-86. doi: 10.3758/bf03196772. PMID 16523997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Different Mixed Condition (DM) | Different Single Condition (DS) | Same Task (ST) Practice Control | Non-WM Placebo Control (PC)
Started | 21 | 25 | 22 | 22
Completed | 19 | 22 | 21 | 18
Not Completed | 2 | 3 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Different Mixed Condition (DM) | Different Single Condition (DS) | Same Task (ST) Practice Control | Non-WM Placebo Control (PC) | Total
Number analyzed (Participants) | 21 | 25 | 22 | 22 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 6 | 4 | 12
  >=65 years | 20 | 24 | 16 | 18 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.95 (6.34) | 72.56 (6.32) | 71.36 (7.82) | 70.77 (6.76) | 71.92 (6.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 14 | 18 | 68
  Male | 5 | 5 | 8 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 20 | 24 | 21 | 22 | 87
  Unknown or Not Reported | 00 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 20 | 22 | 20 | 22 | 84
  More than one race | 0 | 1 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 25 | 22 | 22 | 90
Working Memory Composite [Mean (Standard Deviation); unit: z-score] — Mean z-score of five measures of working memory: Lexical Decision Span, Category Span, Reading Span, Operation Span, and Count Span (e.g., Conway et al., 2005). Higher scores indicate better performance. A z-score of 0 represents the sample mean; units are the standard deviations of the sample (e.g., a score 0.5 would indicate that mean for the group was a half standard deviation above the mean of the entire sample). Clinically relevant scores are unknown.
  z-score | 0.10 (0.86) | -0.05 (0.77) | -0.01 (0.91) | -0.12 (0.55) | -0.02 (0.77)
Education Level [Mean (Standard Deviation); unit: years] — Number of years of formal education (12=high school diploma or GED; 16=completed college; 18=master's degree 20=advanced degree)
  years | 16.29 (2.10) | 16.84 (2.21) | 16.46 (1.84) | 15.93 (2.17) | 16.39 (2.08)

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Working Memory
Description: Average change in working memory from pre- to posttest in z-score units ("standard unit change"). For each working memory measure (Reading Span, Lexical Decision Span, Category Span, Operation Span, and Count Span), the change in z-score units was calculated [(posttest score - pretest score) / standard deviation of the scores at pretest)]. The score reported is the mean of these 5 values. A z-score of 0 represents no change from pretest to posttest; the unit is the standard deviations of the sample at pretest (e.g., a score 0.5 would indicate a half standard deviation improvement in overall working memory). There is no agreed upon standard of clinical significance for improvement in working memory
Time Frame: Change from baseline to 5-6 wks after pretest
Population: Numbers of participants (N=80) differ from baseline (N=90) because 10 participants declined to continue the research activities.
Measure: Mean (Standard Deviation); unit: Standard unit change
Arm/Group | Different Mixed Condition (DM) | Different Single Condition (DS) | Same Task (ST) Practice Control | Non-WM Placebo Control (PC)
Number analyzed (Participants) | 19 | 22 | 21 | 18
Standard unit change | 0.42 (1.40) | 0.26 (0.66) | -0.01 (0.57) | 0.04 (0.38)
Statistical Analysis 1: Comparison: Different Mixed Condition (DM) vs Different Single Condition (DS) vs Same Task (ST) Practice Control vs Non-WM Placebo Control (PC); Test type: Superiority; p = 0.355, ANOVA; Mean Difference (Final Values) = 0.38

2. Primary Outcome: Change in Reading Span
Description: Change in Reading Span score from pre- to posttest in z-score units ("standard unit change"). The change in z-score units was calculated [(posttest score - pretest score) / standard deviation of the scores at pretest)]. A z-score of 0 represents no change from pretest to posttest; the unit is the standard deviations of the sample at pretest (e.g., a score 0.5 would indicate a half standard deviation improvement in overall working memory). There is no agreed upon standard of clinical significance for improvement in working memory
Time Frame: Change from Baseline to 5-6 weeks after pretest
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard unit change
Arm/Group | Different Mixed Condition (DM) | Different Single Condition (DS) | Same Task (ST) Practice Control | Non-WM Placebo Control (PC)
Number analyzed (Participants) | 21 | 22 | 21 | 18
standard unit change | 0.70 (0.66) | 0.06 (0.85) | -0.03 (0.77) | 0.14 (0.66)
Statistical Analysis 1: Comparison: Different Mixed Condition (DM) vs Different Single Condition (DS) vs Same Task (ST) Practice Control vs Non-WM Placebo Control (PC); Test type: Superiority; p < .02, ANOVA; Mean Difference (Final Values) = 0.56 — This is the difference between the Different Mixed and Placebo Control conditions

3. Secondary Outcome: Training Gains on the Reading Span Task in Phase 2
Description: In Phase 2, training data on the target task (Reading Span) is collected over 10 days. Training gains are estimated by the coefficients for the condition contrast by training interaction in a linear mixed effects model, in which mean working memory score across training days was modeled as a function of the Phase 1 training condition. Using the lme4 and lmerTest packages for R version 4.2.2, a mixed-effects linear regression model was employed to model the mean daily span score with condition and training day as the fixed factors, and a by-subject random intercept, using the restricted maximum likelihood (REML) method of estimation.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: coefficient
Arm/Group | Different Mixed Condition (DM) | Different Single Condition (DS) | Same Task (ST) Practice Control | Non-WM Placebo Control (PC)
Number analyzed (Participants) | 19 | 21 | 20 | 17
coefficient | .021 (.011) | .034 (.010) | .021 (.010) | 0 (0)
Statistical Analysis 1: Comparison: Different Mixed Condition (DM) vs Different Single Condition (DS) vs Same Task (ST) Practice Control vs Non-WM Placebo Control (PC); Test type: Other; p < .05, Mixed Models Analysis — for contrasts of DM, DS, and ST groups relative to the PC group

ADVERSE EVENTS:
Time Frame: 6 to 8 weeks
Arm/Group | Different Mixed Condition (DM) | Different Single Condition (DS) | Same Task (ST) Practice Control | Non-WM Placebo Control (PC)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/25 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/25 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/25 | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT05672771/Prot_SAP_ICF_000.pdf